CLINICAL TRIAL: NCT02938832
Title: The CardioDiet Trial
Brief Title: Does the Advice to Eat a Mediterranean Diet With Low Carbohydrate Intake, Compared With a Low-fat Diet, Reduce Diabetes and Cardiovascular Disease?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Fredrik H Nystrom, Professor, MD, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CardioDiet
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Ischemic Heart Disease
Keywords: cardiovascular disease, diet, diabetes
MeSH Terms: conditions — Myocardial Ischemia; Cardiovascular Diseases; Diabetes Mellitus | interventions — Eating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional low-fat diet advice (Active Comparator): Advice on traditional low-fat diet by dietician
  Interventions: Behavioral: Advice on what food to choose and eat
- Mediterranean diet advice (Active Comparator): Advice on a Mediterranean dietary regime with reduced carbohydrates
  Interventions: Behavioral: Advice on what food to choose and eat

INTERVENTIONS:
Behavioral: Advice on what food to choose and eat — Dietary advice

SUMMARY:
This is a multi-centre, open, randomised study in patients treated for ischemic heart disease in Linköping, Norrköping and Jönköping hospitals. One thousand two hundred patients who are treated at the cardiac rehabilitation units will be consecutively recruited during three years. The patients will be randomised 1:1 to be given advice on a 1) Mediterranean diet with an energy content (E%) from carbohydrates between 25-30% or to 2) a traditional low-fat diet with 45-60 E% from carbohydrates. All eligible patients will be asked if they want to participate and provided with written information about the study when they are discharged from the hospital after treatment for ischemic heart disease. The decision to participate or not will be given at the following outpatient treatment at the cardiac rehabilitation unit. When the signed informed consent to participate in the study has been provided, the patient will be randomised to advice of either of the two dietary regimes.

DETAILED DESCRIPTION:
Aim To compare advice on a Mediterranean diet with an energy content (E%) from carbohydrates between 25-30 E% with a traditional low-fat diet with 45-60 E% from carbohydrates.

Primary outcome Incidence of diabetes in non-diabetic patients or glycaemic control in patients with known diabetes.

Secondary outcome Recurrence of cardiovascular disease, blood lipid levels, quality of life by questionnaires.

Study design and study population This is a multi-centre, open, randomised study in patients treated for ischemic heart disease in Linköping, Norrköping and Jönköping hospitals. One thousand two hundred patients who are treated at the cardiac rehabilitation units will be consecutively recruited during three years. The patients will be randomised 1:1 to be given advice on a 1) Mediterranean diet with an energy content (E%) from carbohydrates between 25-30% or to 2) a traditional low-fat diet with 45-60 E% from carbohydrates. All eligible patients will be asked if they want to participate and provided with written information about the study when they are discharged from the hospital after treatment for ischemic heart disease. The decision to participate or not will be given at the following outpatient treatment at the cardiac rehabilitation unit. When the signed informed consent to participate in the study has been provided, the patient will be randomised to advice of either of the two dietary regimes.

ELIGIBILITY:
Inclusion Criteria: Patients treated for ischemic heart disease who are followed up at the cardiac rehabilitation units

Exclusion Criteria: Inability to affect food choice. Severe concomitant disease such as malignancy, renal failure, heart failure or psychiatric disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2016-10; Primary Completion 2021-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Diabetes incidence | 3 years
  Hba1c > 48 mmol/mol

SECONDARY OUTCOMES:
Cardiovascular disease | 3 years and more
  CVD incidence based on national registries
Quality of Life | 3 years
  QoL by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik H Nystrom, MD professor, Principal Investigator — Faculty of Medicine and Health Sciences, Linköping University
Locations (1):
- University Hospital of Linkoping, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes